CLINICAL TRIAL: NCT07406880
Title: Positive Psychology-Based Ecological Momentary Intervention for Well-Being in College Students: A Randomized Controlled Trial
Brief Title: Positive Psychology - Based EMl for Enhancing Well-Being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSEARS20231201008-03
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants Study

STUDY DESIGN:
Intervention Model Description: This three-arm randomized controlled trial evaluates a 14-day Positive Psychology- based Ecological Momentary Intervention (EMI). All participants complete twice-daily assessments of emotions and activities, as well as a Daily Diary at 9:00 PM each day. Participants are randomly assigned to one of three groups: 1. EMI Group: Receives algorithm triggered positive psychology exercises (e.g., gratitude, mindfulness) when their real-time emotional states fall below a predefined threshold. 2. Active Control Group: Completes the same set of exercises on a fixed schedule, regardless of momentary emotional state. 3. No-Intervention Control Group: Completes all assessments but receives no intervention exercises.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMI Group (Experimental): Participants in this group will use the app which delivers EMI exercises adaptively. Twice daily, the app assesses their momentary affect and well-being. If scores fall below a preset threshold, a corresponding intervention exercise (e.g., gratitude, mindfulness) is automatically triggered. They also complete a daily evening assessment. The intervention lasts 14 days.
  Interventions: Behavioral: Ecological Momentary Intervention
- Active Control Group (Active Comparator): Participants in this group will use the app to complete a fixed set of six EMI exercises twice daily, regardless of their current emotional state. This controls for the general effect of receiving the intervention content and frequency. They also complete the same daily evening assessment as the other groups. The phase lasts 14 days.
  Interventions: Behavioral: Active Control
- No-Intervention Control Group (No Intervention): Participants in this group will use the app only for assessment purposes. They complete the same twice-daily momentary assessments and the daily evening assessment as the other groups, but do not receive any intervention exercises. This controls for the effects of repeated self-monitoring. The phase lasts 14 days.

INTERVENTIONS:
Behavioral: Ecological Momentary Intervention — This is a smartphone-based ecological momentary intervention (EMI) that delivers psychological exercises (e.g., gratitude, mindfulness) in an adaptive, "as-needed" manner. Twice daily, the app algorithm assesses a participant's self-reported momentary affect and well-being. If the scores fall below a preset, moderate threshold, a corresponding intervention exercise is automatically triggered. The goal is to provide personalized support at moments of greatest need.
  Arms: EMI Group
Behavioral: Active Control — This is a smartphone-based ecological momentary intervention (EMI) that delivers the same suite of psychological exercises on a fixed schedule, regardless of the user's current state. Participants are prompted to complete all six available exercises twice daily. This intervention controls for the general effects of exposure to the exercise content and engagement with the app, allowing for a comparison with the adaptive, algorithm-guided EMI.
  Arms: Active Control Group

SUMMARY:
This study aims to evaluate the acceptability and effectiveness of a positive psychology-based ecological momentary intervention (EMI) for enhancing well-being in college students. A three-arm randomized controlled trial (RCT) will assess the impact of a dynamic EMI that delivers personalized exercises when participants' real-time affect or well-being scores fall below a predefined threshold, compared to control conditions. Primary outcomes include changes in well-being and mental health, evaluated through a mixed-methods approach combining quantitative measures and qualitative interviews.

DETAILED DESCRIPTION:
This study aims to evaluate a Positive Psychology-based Ecological Momentary Intervention (EMI) designed to enhance well-being among college students. A three-arm randomized controlled trial (RCT) will be conducted to examine the intervention's effectiveness. The EMI integrates core positive psychology practices-such as gratitude, mindfulness, and acts of kindness-and is delivered through a mobile application in real time. The intervention features a dynamic, adaptive algorithm that provides personalized exercises when participants' real-time affect or well-being scores fall below a predefined threshold. Primary outcomes include changes in well-being and mental health . A mixed-methods design will be employed, combining quantitative assessments at baseline, post-intervention, and one-month follow-up with qualitative post-intervention interviews to gain an in-depth understanding of the intervention's impact and user experience.

ELIGIBILITY:
Inclusion Criteria:

* Participants in our study are healthy college students.
* Have smartphone, and have access to the internet.

Exclusion Criteria:

* Unable to use a smartphone.
* Have significant cognitive impairment that prevents participation in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Affect | Baseline (pre-intervention); Immediately after the intervention (2 week after baseline)); 1-month follow-up (1 month after intervention)
  The 20-item Positive and Negative Affect Schedule Short Form (PANAS-SF) will be used to measure affective states. This scale comprises two subscales: Positive Affect (10 items) and Negative Affect (10 items). Each item is rated on a 5-point scale from 1 (very slightly or not at all) to 5 (extremely). Higher scores on each subscale indicate higher levels of the respective affect.
Happiness | Baseline (pre-intervention); Immediately after the intervention (2 weeks after baseline); 1-month follow-up (1 month after intervention)
  The 4-item Subjective Happiness Scale (SHS) will be utilized to assess participants' subjective happiness. Each item will be rated on a 7-point Likert scale. Elevated scores on the scale indicate a greater level of subjective happiness.
Flourishing | Baseline (pre-intervention); Immediately after the intervention (2 weeks after baseline); 1-month follow-up (1 month after intervention)
  The 8-item Flourishing Scale (FS) will be used to measure psychological well-being and self-perceived success in important areas such as relationships, self-esteem, and purpose. Each item is rated on a 7-point scale from 1 (strongly disagree) to 7 (strongly agree), with higher scores indicating a greater level of psychological well-being.
Satisfaction with Life | Baseline (pre-intervention); Immediately after the intervention (2 weeks after baseline); 1-month follow-up (1 month after intervention)
  Satisfaction with life is measured by the 5-item Satisfaction with Life Scale (SWLS). All items are rated on a 7-point scale from 1 (strongly disagree) to 7 (strongly agree), with higher scores indicating higher satisfaction with life.
Psychological distress | Baseline (pre-intervention); Immediately after the intervention (2 weeks after baseline); 1-month follow-up (1 month after intervention
  The 21-item Depression Anxiety Stress Scale (DASS-21) will be used to measure the negative emotional states of depression, anxiety, and stress. Each subscale contains 7 items, rated on a 4-point severity scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Higher scores indicate more severe levels of depression, anxiety, or stress.

SECONDARY OUTCOMES:
State Subjective Happiness | During the 14-day intervention period, this measurement is conducted twice per day as part of the momentary assessments, and once each evening as part of the Daily Diary assessment at 9:00 PM.
  State Subjective Happiness will be measured by the 2-item Subjective Happiness Scale with each item rated on a 7-point Likert scale from 1 (not a very happy person) to 7 (a very happy person).
State affect | During the 14-day intervention period, this measurement is conducted twice per day as part of the momentary assessments, and once each evening as part of the Daily Diary assessment at 9:00 PM.
  State affect will be tapped by the 9-item Ecological Mood Indicator. Participants indicate their momentary feelings on a 7-point Likert scale ranging from 1 (not at all) to 7 (extremely), for NA (e.g., depressed, worried/anxious, and unhappy) and PA (e.g., joyful, happy, and enjoyment/fun)
State Well-Being | During the 14-day intervention period, this measure is also administered each evening at 9:00 PM as part of the Daily Diary assessment.
  State stress will be measured with one item adapted from the Psychological Stress Measure (PSM-9) using a 5-point Likert scale ranging from 0 (Not at all stressed) to 4 (Extremely stressed).
State Anxiety and Depression | During the 14-day intervention period, this measure is also administered each evening at 9:00 PM as part of the Daily Diary assessment.
  State Anxiety and Depression will be measured with the four-item Patient Health Questionnaire for Depression and Anxiety (PHQ-4). Responses are scored as 0 ("not at all"), 1 ("several days"), 2 ("more than half the days"), or 3 ("nearly every day"), with the total score on this composite measure ranging from 0 to 12.
State Stress | During the 14-day intervention period, this measure is also administered each evening at 9:00 PM as part of the Daily Diary assessment.
  State stress will be measured by a single item asking participants to rate their current stress level on a 5-point Likert scale ranging from 0 (Not at all stressed) to 4 (Extremely stressed).

OTHER OUTCOMES:
Socio-demographic variables | Baseline (pre-intervention)
  The following socio-demographic variables such as sex, age, grade, and family income will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong